CLINICAL TRIAL: NCT03434782
Title: Effect of Low-level Light Therapy Associated With Potassium Nitrate in the Control of Post-bleaching Dental Sensitivity: a Randomized, Double-blind, Split-mouth, Controlled Trial
Brief Title: Effect of Laser and Potassium Nitrate Application on the Sensitivity Control in Bleached Teeth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Cecy Martins Silva, Associate Professor, Universidade Federal do Para
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UFPara-002
Record Dates: First submitted 2018-01-16; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Hydrogen Peroxide; Low-Level Light Therapy; potassium nitrate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- G1- Negative Control (Experimental): Group with no desensitizing treatment. Prior to bleaching therapy, a water-soluble placebo gel, with non-active agent will be applied to dental vestibular surfaces. After bleaching therapy, the LASER tip will be positioned in two points (apical and cervical), without light emission (placebo).
  Interventions: Drug: In-office dental bleaching
- G2- LASER (Positive Control) (Experimental): Group treated with placebo gel before bleaching and with LLLT after in-office bleaching.
  Interventions: Drug: In-office dental bleaching; Drug: Low Level Laser Therapy
- G3- KNO3 (Positive Control) (Experimental): Group treated with desensitizing gel before bleaching and after in-office bleaching, the LASER tip will be positioned in two points (apical and cervical), without light emission (placebo).
  Interventions: Drug: In-office dental bleaching; Drug: 5% potassium nitrate / 2% sodium fluoride gel
- G4- KNO3 + LASER (Experimental): Group treated with desensitizing gel before bleaching and with LLLT after in-office bleaching.
  Interventions: Drug: In-office dental bleaching; Drug: Low Level Laser Therapy; Drug: 5% potassium nitrate / 2% sodium fluoride gel

INTERVENTIONS:
Drug: In-office dental bleaching — The group will receive in-office bleaching treatment. Three 15-minute applications of the 35% hydrogen peroxide gel were performed, totaling 45 minutes in each of the 3 sessions, with a 7-day interval.
  Other Names: 35% hydrogen peroxide
Drug: Low Level Laser Therapy — It will be used the infrared spectrum with wavelength of 808 nm in its active environment AsGaAl, in two points: cervical and apical region of the incisors, canines and premolars.
  Other Names: LLLT
  Arms: G2- LASER (Positive Control); G4- KNO3 + LASER
Drug: 5% potassium nitrate / 2% sodium fluoride gel — 5% potassium nitrate / 2% sodium fluoride gel will be applied for 10 minutes on the vestibular surface of all pre-bleached dental elements, following the manufacturer's protocol.
  Other Names: desensitizing therapy
  Arms: G3- KNO3 (Positive Control); G4- KNO3 + LASER

SUMMARY:
To investigate the effects of desensitizing agents on the dental bleaching process, testing the hypothesis that they may control dental sensitivity.

DETAILED DESCRIPTION:
The objective of this double blind, randomized and controlled clinical study, was to evaluate the efficacy of potassium nitrate / sodium fluoride (KNO3 / KF) gel associated with LLLT (Low Level Light Therapy) on teeth that were exposed to 35% hydrogen peroxide during 3 weeks of bleaching treatment. Methods: 50 volunteers were evaluated through the split-mouth model, where the hemiarcates were randomized and later allocated in one of the experimental groups: G1 (negative control)- group with no desensitizing treatment, only bleached; G2 (positive control)- group treated with LLLT + placebo gel; G3- group treated with placebo laser application + 5% KNO3 / 2% KF gel; and G4- group treated with LLLT + 5% KNO3 / 2% KF gel.

ELIGIBILITY:
Inclusion Criteria:

* Absence of active carious lesions;
* Never undergone bleaching therapy;
* Good oral hygiene;
* Do not present hypersensitivity;
* Do not smoke;
* Not being pregnant;
* Presence of at least 28 teeth in oral cavity.

Exclusion Criteria:

* Presence of periodontal disease;
* Presence of cracks or fractures;
* Presence of restorations and prostheses;
* Presence of gastroesophageal dysfunction;
* Patients with severe internal dental dimming;
* Presence of periodontal disease;
* Presence of dentin exposure in anterior and/or posterior teeth.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Stimulated pain intensity in different assessment times (P15) | 15 days, with assessments in the 1st, 8th and 15th day of the treatment
  The stimulated pain intensity was self reported by the patients with a modified visual analog scale, from 0 to 3, where 0 means "no pain", 1 is "mild pain", 2 is "moderate pain" and 3 is "severe pain". For all groups, the patients evaluated the stimulated pain intensity two times per session: before and after the treatment in the same day. Thus, in total each patient reported the pain intensity 6 times, two times in the first day (1st session), two times in the eighth day (2nd session) and two times in the fifteenth day (3rd session).

SECONDARY OUTCOMES:
Non-stimulated pain intensity measure, (P21) | 21 days
  Self reported non-stimulated pain intensity was assessed daily, during 21 days, through self-perception questionnaire, answered by the patients from the first tooth bleaching session until one week after the last session. The evaluation was performed by each patient, according to a modified visual analog scale, as follows: 0- no pain, 1 mild pain, 2 - moderate pain and 3 -severe pain

CONTACTS AND LOCATIONS:
Locations (1):
- Brennda Lucy Freitas de Paula, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reis A, Dalanhol AP, Cunha TS, Kossatz S, Loguercio AD. Assessment of tooth sensitivity using a desensitizer before light-activated bleaching. Oper Dent. 2011 Jan-Feb;36(1):12-7. doi: 10.2341/10-148-CR. Epub 2011 Mar 24. PMID 21488723
- [Result] Moosavi H, Arjmand N, Ahrari F, Zakeri M, Maleknejad F. Effect of low-level laser therapy on tooth sensitivity induced by in-office bleaching. Lasers Med Sci. 2016 May;31(4):713-9. doi: 10.1007/s10103-016-1913-z. Epub 2016 Mar 10. PMID 26964798
- Available data/document: Study Protocol: 60622416.1.0000.0018 — http://aplicacao.saude.gov.br/plataformabrasil/visao/pesquisador/gerirPesquisa/gerirPesquisaAgrupador.jsf